CLINICAL TRIAL: NCT00961727
Title: Implementation of Bedside PEWS at Credit Valley Hospital
Brief Title: Implementation of Bedside Pediatric Early Warning Systems (PEWS)
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Christopher Parshuram, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000009778
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Clinically Deteriorating Paediatric Patients
Keywords: Bedside Pews; Credit Valley Hospital; The Bedside Paediatric Early Warning System; clinically deteriorating

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PEWS System of Care
  Interventions: Other: Bedside Paediatric Early Warning System (Bedside PEWS)

INTERVENTIONS:
Other: Bedside Paediatric Early Warning System (Bedside PEWS) — The Bedside PEWS is comprised of 4 components; [1] an expert derived, multi-centre validated severity of illness score, [2] an inter-professionally developed documentation record into which the severity of illness score is embedded, [3] a series of score-matched care recommendations based on the opinions of over 280 paediatric health care professionals, and [4] an educator-developed education-implementation program.

SUMMARY:
Timely identification, referral and treatment of children who are clinically deteriorating while admitted to hospital wards is a fundamental element of inpatient care. In community hospitals, advantages including greater continuity of inpatient-outpatient care, improved geographic access for families, and lower healthcare system costs, may be undermined if children with evolving critical illness are not recognized and transferred in a timely manner. The Bedside Paediatric Early Warning System (Bedside PEWS) is a system of care designed to augment existing expertise and to provide a safety net for children who are clinically deteriorating while admitted to hospital wards. The Bedside PEWS is comprised of 4 components; [1] an expert derived, multi-centre validated severity of illness score, [2] an inter-professionally developed documentation record into which the severity of illness score is embedded, [3] a series of score-matched care recommendations based on the opinions of over 280 paediatric health care professionals, and [4] an educator-developed education-implementation program.

DETAILED DESCRIPTION:
We will be performing a prospective observational study of care outcomes, physician workload and frontline staff perceptions before and after the implementation of Bedside PEWS in a community paediatric hospital. We plan to evaluate the outcomes of patients who were admitted to the 22-bed paediatric inpatient unit and were less than 18 years of age at hospital admission, and the healthcare professionals caring for them during their inpatient stay.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the paediatric inpatient unit at Credit Valley Hospital from June 2008-December 2008

Exclusion Criteria:

* Patients over 18 years of age

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients admitted to the 22-bed paediatric inpatient unit and were less than 18 years of age at hospital admission
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Significant clinical deterioration events | -3 months, +2months, and+5months after implementation

SECONDARY OUTCOMES:
'stat' calls to the paediatrician | 3 months before and 5 months after implementation
'stat' calls to the respiratory therapist | 3 months before and 5 months after implementation
immediate calls to treat near or actual cardiopulmonary arrest - 'code-blue' | 3 months before and 5 months after implementation

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Parshuram, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada